CLINICAL TRIAL: NCT06101368
Title: Effect of Physical Activity on Neurogenesis in Peripheral Diabetic Neuropathy Type-II Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Dr Danish Raouf, Physical Therapist, Health Education Research Foundation (HERF)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RHS/EC/02-06-2023-011
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Type II Diabetes Mellitus With Neurological Manifestations
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Combined Aerobic and Resistance Training) (Experimental): Group A will perform aerobic and resistance exercises at a moderate level. Brisk Walk on treadmill 5 days/week with 40-70% of Vo2max (maximal aerobic capacity) 150 min/week 50-55% humidity and a room temperature of 24-25 °C will maintain. The subject will wear insole proper fitted shoes. Aerobic exercise will be conducted for a total of 30 minutes per session for 5 days for 12 weeks. This protocol will be followed by a 10-minute warm-up and cool-down. Followed by 10-15 minutes of resistance-based exercises at a moderate intensity of three sets with 15 repetitions of upper and lower limbs respectively i.e. Dumbbell biceps curl, Standing dumbbell triceps extension, Dumbbell stiff-legged deadlifts and Dumbbell squats Resistance loads will be 40-50% of one repetition maximum. The resting interval between resistance training sets will be < 1 min.
  Interventions: Behavioral: Phsical Activity
- Control Group (Other): The control group will maintain their usual activity level, foot care, diet, and blood glucose diary on a regular basis. Continue the prescribed medication
  Interventions: Drug: Medication

INTERVENTIONS:
Behavioral: Phsical Activity — Combined Aerobic and Resistance Training
  Arms: Physical Activity (Combined Aerobic and Resistance Training)
Drug: Medication — The drug will maintain their usual activity level, foot care, diet, and blood glucose diary on a regular basis. Continue the prescribed medication
  Arms: Control Group

SUMMARY:
Approximately 425 million people worldwide suffer from diabetes, making it a global epidemic. Diabetes consumes 12% of the global health budget, addressing the disease and its complications. In Pakistan, the estimated prevalence of diabetes stands at 9.8%, affecting both males and females. Diabetic peripheral neuropathy is a common complaint that significantly impacts patients' quality of life. Neuropathy is prevalent in 40-55% of diabetes cases, and its incidence rises with age. Additionally, exercise can promote neurogenesis and the release of beneficial factors like BDNF, contributing to improved cognitive function and mood. Aerobic exercises are recommended for managing type 2 diabetes, while resistance training can improve glycemic control and muscle health. Further research is needed to understand the effects of physical activity on neurogenesis in diabetic peripheral neuropathy patients and gender-specific influences on glucose metabolism. The study aims to enhance peripheral neurogenesis, glycemic control, and sensory functions, ultimately improving the overall quality of life for patients.

DETAILED DESCRIPTION:
The study design is a randomized controlled trial, and participants will be blinded to avoid interaction. A convenience sampling technique will be used, and the study will take place at Pakistan Railways Hospital and Quaid-E-Azam University. It will span two years after receiving approval. Inclusion criteria specify the type of patients eligible for the study, while exclusion criteria identify conditions that disqualify participants. Various data collection tools and tests will be used, including Neuropathy Total Symptom Scale (NTSS-6), Berg Balance Scale, HbA1c, nerve conduction studies, blood glucose level measurements, dynamometer, and questionnaires assessing quality of life.

The study procedure involves participant recruitment, randomization into treatment and control groups, baseline assessments, and a 12-week intervention for the treatment group. This includes both aerobic exercise (treadmill) and resistance training for the lower and upper extremities. Control group participants will continue their regular medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type-II Peripheral Diabetic Neuropathy
* Neuropathy Total Symptom Scale (NTSS-6)>6
* loss of protective sensation to detect a 10-gram Semmes Weinstein Monofilament on either foot at one of four sites tested or a vibration perception threshold value of 25V or more at either foot's hallux
* Numbness or reduced ability to feel pain or temperature changes.
* Able to Perform 20 minutes per week >2 bouts of physical activity
* Tingling or burning sensation.
* Sharp pains or cramps.
* Increased sensitivity to touch
* Symptoms last ≥ 6 months
* HbA1c above 6.5% <12%
* Berg Balance Scale score 45-56

Exclusion Criteria:

* Patients with walking difficulty
* Retinopathy & poor vision
* Inability to engage in activity without assistance
* Peripheral vascular disease e.g. ABI <0.6
* orthostatic hypotension, resting heart rate above 100 bpm any Cardiac Issues
* Any diagnosed neuro-psychological issue e.g. depression, dementia or anxiety
* Lower limb amputation,foot deformity or ulceration
* Acute injury
* Hip and Knee OA

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Brain Derived Neurotrophic Factor (BDNF) | Baseline to after 12th Week
  BDNF is a member of the trophic factors of nerve regeneration microenvironment and therefore involved in the regulation of nerve fiber regeneration and protection of neurons
Nerve Growth Factor (NGF) | Baseline to after 12th Week
  Nerve growth factor (NGF) is a neurotrophic protein essential for the growth, differentiation, and survival of sympathetic and sensory afferent neurons during development
Vascular Endothelial Growth Factor (VEGF) | Baseline to after 12th Week
  VEGF enhances nerve blood flow and oxygen supply by inducing angiogenesis, in response to nerve ischemia and hypoxia caused by Diabetic Periphral Neuropathy
HBA1c | Baseline to after 12th Week
  HbA1c levels are associated with increased severity of peripheral neuropathy in patients with diabetes mellitus.
Nerve Conduction Study (NCS) | Baseline to after 12th Week
  A nerve conduction study (NCS) can quantitatively detect peripheral nerve dysfunction, even in the pre-symptomatic stage of DPN onset.
Berg Balance scale (BBS) | Baseline, after 4th week, after 8th week and after 12th week
  The Berg Balance Scale (BBS) is a widely used clinical assessment tool that measures an individual's static and dynamic balance abilities. It is not specific to diabetic neuropathy but can be used to assess balance in individuals with various neurological and musculoskeletal conditions, including diabetic neuropathy.
Neuropathy Total Symptom Scale (NTSS-6) | Baseline, after 4th week, after 8th week and after 12th week
  Neuropathy Total Symptom Score-6 Questionnaire (NTSS-6) is a valid instrument for assessing the positive symptoms of diabetic peripheral neuropathy (DPN). Graphic representation of pain.
Dynamometry lower limb | Baseline, after 4th week, after 8th week and after 12th week
  Dynamometry is a method used to measure muscle strength, and it can be particularly useful in assessing muscle strength in the lower limbs of individuals with diabetic neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar A Awan, PhD, Principal Investigator — Health Education Research Foundation; Raheela Kanwal, PhD, Principal Investigator — College of Applied Medical Sciences, University of Hail, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided